CLINICAL TRIAL: NCT07079501
Title: 8-week Efficacy Clinical Study on Chinese Healthy Female, 40 Subjects
Brief Title: Eye Cream 8-Week Efficacy Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25005004
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Wrinkles and Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Eye Cream Arm (Experimental): Participants will apply the test eye cream (Formula# 899675 44A) twice daily on full face and neck for 8 weeks. The study is designed to evaluate improvements in facial wrinkles, eye bags, dark circles, skin firmness, elasticity, radiance, and smoothness in healthy Chinese women aged 20-50.
  Interventions: Other: Test Eye Cream (Formula# 899675 44A)

INTERVENTIONS:
Other: Test Eye Cream (Formula# 899675 44A) — A white cream formulated as eye cream (Formula# 899675 44A) provided by L'Oréal R&I China. Participants will apply 1ml of the product on the full face and neck twice daily for 8 weeks. The aim is to evaluate its efficacy on facial wrinkles, eye bags, dark circles, and other skin aging signs in healthy Chinese women.

SUMMARY:
To investigate efficacy on test cream [Formula#899675 44A] on female subjects after 2-week wash-out and 8-week repeated application.

50 female adult subjects will be enrolled in the study, recruited according to inclusion and non-inclusion criteria listed above. At least 40 subjects should complete the study in this 10-week study (wash-out phase for 2-week and treatment phase for 8 weeks). Subjects will need to refrain from using any product other than the provided products on face during the study phase.

1. Clinical Assessment (N=40 at least):

   *Clinical scoring for smoothness (visual), elasticity, cheek plumpness, radiance, global fine lines, firmness, dry lines, small folds on nasolabial zone (Atlas), underneath eye wrinkles (Atlas), forehead wrinkles (Atlas), nasolabial fold (Atlas), cheek folds: (Atlas), wrinkles of the corner of the lips (Atlas), inter-ocular wrinkles (Atlas), crow's feet wrinkles (Atlas), glabellar wrinkles (Atlas), horizontal neck fold (Atlas) by Dermatologist at T-2W, T0, Timm, T2W, T4W, T8W.
   * Clinical scoring for eye bag (Atlas), intensity and coverage of dark circle (vascular) (0~4 scale) by Dermatologist at T-2W, T0, T2W, T4W, T8W.
2. Image Capture and Analysis (N=40 at least):

   *The facial photo will be captured by VISIA CRP (Canfield, Gen 5.0) on left, front and right sides with Standard, Cross-polarized, Parallel-Polarized, Primos operated by trained technician at T0, Timm, T2W, T4W, T8W.

   -Demo with mark line for forehead wrinkles, underneath eye wrinkles, crow's feet wrinkles
   * Primos demo for crow's feet wrinkles

   Image Analysis by Primos 5.8E:

   -Wrinkle volume (mm³), Wrinkle area (mm²), total length (mm), count of crow's feet wrinkles

   *The facial photo will be captured by COLORFACE® (Newtone Technologies) on front side with closed eyes under Cross-Polarized mode at T0, T2W, T4W, T8W.
   * Demo with dark circles.

   Image Analysis by Image-Pro Plus 7.0:
   * L*, a*, b* and ITA° focus on underneath eye zone.

     *The local 3D photo will be captured by Primos-lite (Canfield) on both sides of underneath eye zone for eye bags by trained technician at T0, T2W, T4W, T8W. (at least 10 subjects with eye bags (Altas, 0~6 scale) grade≥2)
   * Demo with eye bags.

   Image Analysis by Primos 5.8E:

   -Rising Volume (mm³) of eye bags

ELIGIBILITY:
Inclusion Criteria:

Prospective subjects meeting all the criteria below will be eligible for enrolment:

1. Chinese women aged from 20-50 years old (must have subjects aged from 20-30 y.o.).
2. All skin types, with about 50% sensitive skin (self-declared).
3. Regular users of cleanser, anti-aging cream and sunscreen products.
4. Self-claim with wrinkles concern, also with lack of elasticity, firmness and plumpness.
5. Clinical grading by dermatologist on global face following:

   Skin firmness (0-9 scale, 3≤ grade≤ 6) Skin elasticity (0-9 scale, 3≤ grade≤ 6) Skin radiance (0-9 scale, 3≤ grade≤ 6) Skin smoothness (0-9 scale, 3≤ grade≤ 6) Skin plumpness (0-9 scale, 3≤ grade≤ 6)
6. Clinical grading by dermatologist on face following:

   Underneath eye wrinkles (Atlas Page 44~45, 2≤ grade≤ 5) Forehead wrinkles (Atlas Page 30~31, 1<grade≤ 4) Nasolabial folds (Atlas Page 52~53, 1<grade) Crow's feet wrinkle (Atlas Page 36~37, 1<grade) Inter ocular wrinkles (Atlas Page 38~39, 1<grade) Wrinkles of the corner of the lips (Atlas Page 60~61, 1<grade) Dark circle (vascular) (0-4 scale, 2≤ grade) Eye bags (Atlas Page 42-43, 2≤ grade) (at least N=10)
7. No disagreement of dermatologist because of other reasons that exclude the participation of the subject.
8. In general good health at the time of the study.
9. Willing and able to participate as evidenced by signing of informed consent and photo release form.
10. Must be willing to comply with all study protocol requirements (pay attention to: only use the provided product during the study, not take topical or oral treatment like retinol, hormone, anti-oxidant health-care products which may impact the efficacy of study).

Exclusion Criteria:

* 1.Pregnant or breast-feeding woman or woman planning pregnancy during the study.

  2.Subject deprived of rights by a court or administrative order. 3.Major subject to a guardianship order. 4.Subject residing in a health or social care establishment. 5.Patient in an emergency setting. 6.Subject with a skin disease in the test areas (particularly e.g, acne, rosacea, eczema).

  7.Subjects with history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, medication, cosmetic or personal care products or ingredients.

  8.Subject presenting a stable or progressive serious disease (per investigator's assessment).

  9.Immuno-compromised subject. 10.Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).

  11.Subjects regularly practicing aquatic or nautical sports. 12.Subjects regularly attending a sauna. 13.Subject with cardiovascular or circulatory history. 14.Subject with a history of skin cancer or malignant melanoma. 15.Anti-aging medical beauty project or anti-aging cosmetics clinical research in the last 6 months before study.

  16.Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants in the last 6 months before study.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-11-17 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Change in wrinkle severity score assessed by dermatologist using Skin Aging Atlas | Baseline (T0), Day 14 (T2W), Day 28 (T4W), and Day 56 (T8W)
  Clinical evaluation of facial wrinkles including crow's feet, forehead wrinkles, glabellar lines, nasolabial folds, and eye wrinkles using the Skin Aging Atlas (0-9 scale), conducted by a dermatologist.

SECONDARY OUTCOMES:
Change in skin firmness score (Griffiths scale) | Baseline (T0), Day 14 (T2W), Day 28 (T4W), and Day 56 (T8W)
  Dermatologist grading of skin elasticity using a modified Griffiths scale (0-9), based on tactile skin rebound assessment.
Change in skin elasticity score (Griffiths scale) | Baseline (T0), Day 14 (T2W), Day 28 (T4W), and Day 56 (T8W)
  Dermatologist grading of skin elasticity using a modified Griffiths scale (0-9), based on tactile skin rebound assessment.
Change in skin smoothness score (Griffiths scale) | Baseline (T0), Day 14 (T2W), Day 28 (T4W), and Day 56 (T8W)
  Dermatologist evaluation of skin smoothness using a 0-9 modified Griffiths scale based on visual observation and tactile texture.
Change in skin plumpness score (Griffiths scale) | Baseline (T0), Day 14 (T2W), Day 28 (T4W), and Day 56 (T8W)
  Dermatologist evaluation of skin radiance based on facial glow and uniformity, scored using a modified Griffiths 0-9 scale.
Change in crow's feet wrinkle volume (mm³) | Baseline (T0), Day 14 (T2W), Day 28 (T4W), Day 56 (T8W)
  Quantitative evaluation of wrinkle volume using Primos 5.8 3D imaging system. Measurement includes wrinkle volume (mm³) in the crow's feet region.
Change in crow's feet wrinkle area (mm²) | Baseline (T0), Day 14 (T2W), Day 28 (T4W), Day 56 (T8W)
  Quantitative evaluation of wrinkle area using Primos 5.8 3D imaging. Area (mm²) of the crow's feet region analyzed.
Change in crow's feet wrinkle count | Baseline (T0), Day 14 (T2W), Day 28 (T4W), Day 56 (T8W)
  Counting of visible crow's feet wrinkles using Primos 5.8 system under standardized imaging conditions.
Change in under-eye dark circle pigmentation (L*, a*, b*, ITA° values) | Baseline (T0), Day 14 (T2W), Day 28 (T4W), Day 56 (T8W)
  Colorface® and Image-Pro Plus 7.0 analysis of pigmentation under cross-polarized light. Parameters include L*, a*, b*, and ITA° in the under-eye zone.
Change in eye bag volume (mm³) | Baseline (T0), Day 14 (T2W), Day 28 (T4W), Day 56 (T8W)
  3D volume assessment of under-eye bags using Primos imaging, reported in mm³. At least 10 participants must present with baseline eye bag score ≥2.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai 200072, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
This Data Sharing Plan (DSP) aims to promote the open exchange and reuse of de-identified individual participant data (IPD) from cosmetic clinical research, including study protocols, case report forms (CRFs), and statistical analysis plans (SAPs). The shared data will be made available through compliant platforms to eligible researchers in dermatology, cosmetic science, and related fields, following ethical principles and data protection regulations. Users must sign a Data Use Agreement (DUA) to ensure data security, privacy protection, and compliance with research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18-Month Duration: The data sharing period starts upon study completion and PRS registration completion.
  Timeline:
  Months 2-3: Data de-identification, metadata preparation, and platform integration.
  Month 4: Official launch of data access.
Access Criteria: Primary Platform:
  ResMan (www.medresman.org.cn) - China's leading medical research data repository.
  Eligibility:
  Researchers/affiliates from academic institutions, hospitals, or registered research organizations.
  Engaged in dermatology, cosmetic science, or related fields. Able to demonstrate ethical compliance and data security capabilities.
URL: http://www.medresman.org.cn